CLINICAL TRIAL: NCT07262918
Title: The Impact of Medical TV Drama in Improving Literacy on Asthma: An Online Open-Label Two-arm Randomized Control Trial.
Brief Title: The Impact of Medical TV Drama in Improving Literacy on Asthma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cephas Health Research Initiative Inc, Ibadan, Nigeria (Network)
Responsible Party: Principal Investigator, Emeka Okeke, Director, Cephas Health Research Initiative Inc, Ibadan, Nigeria
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CUL25/0877
Record Dates: First submitted 2025-09-27; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Asthma
Keywords: Asthma; Television; Drama; Literacy; Medical
MeSH Terms: conditions — Asthma; Literacy

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL ARM (NO MEDIAL INTERVENTION) (No Intervention): NO INTERVENTION
- INTERVENTION ARM (MEDIAL INTERVENTION) (Active Comparator): MEDIAL INTERVENTION
  Interventions: Device: TELEVISION DRAMA

INTERVENTIONS:
Device: TELEVISION DRAMA — MEDICAL TV DRAMA
  Arms: INTERVENTION ARM (MEDIAL INTERVENTION)

SUMMARY:
Asthma is an important chronic noncommunicable disease that affects children and adults following a complex immune-mediated mechanism involving airway inflammation, bronchial hyperresponsiveness, and transient and intermittent airway obstruction. A current global empirical study, published in 2025, estimated that asthma affects about 260 million people, and it is responsible for about 455,000 deaths globally. Despite the morbidity and mortality-laden nature of asthma, the awareness and knowledge of this important condition remains low among several populations. Notably, no known multi-country intervention study has ever investigated the effectiveness, acceptability, and usability of medical TV programs in educating young persons on asthma. Therefore, this two-arm randomized control trial (RCT) aims to evaluate the impact of watching a medical TV drama on asthma among a sample of individuals (who do not have prior medical knowledge) from different cultural backgrounds and countries.

DETAILED DESCRIPTION:
Asthma is an important chronic noncommunicable disease that affects children and adults following a complex immune-mediated mechanism involving airway inflammation, bronchial hyperresponsiveness, and transient and intermittent airway obstruction. Asthma is the most common chronic disease in childhood. A current global empirical study, published in 2025, estimated that asthma affects about 260 million people, and it is responsible for about 455,000 deaths globally. Despite the morbidity and mortality-laden nature of asthma, the awareness and knowledge of this important condition remains low among several populations. This knowledge gap can cause poor adherence to treatment. Studies have shown that media entertainment is a potent tool that can be used to deliver complex health information for a desired behavioral change among young people. Therefore, this two-arm randomized control trial (RCT) aims to evaluate the impact of watching a medical TV drama on asthma among a sample of individuals (who do not have prior medical knowledge) from different cultural backgrounds and countries. The insights gained from this online two-arm RCT will contribute to existing knowledge on the area of asthma prevention and control, and it will help to direct policy recommendations for planning health education interventions targeted at young adults.

METHODS Study Design This study will be an online, open-label, parallel-group, two-arm RCT, a rigorous design widely used to evaluate the effectiveness of health interventions. The trial will aim to determine the impact of a medical TV drama episode on asthma-related health literacy among young adults. The design will be informed by evidence suggesting that entertainment media can enhance health knowledge and influence behavior change. Participants will be randomly assigned to either an intervention group (who will view the episode) or a control group (with no exposure), and their knowledge scores will be compared before and after the intervention. The study will follow the CONSORT (Consolidated Standards of Reporting Trials) 2010 guidelines for the reporting of RCTs.

Study Setting and Participants. The trial will be conducted entirely online, a delivery model increasingly adopted for its cost-efficiency, accessibility, and potential to reach a geographically diverse population. Participants will be recruited using social media platforms such as Facebook, Instagram, WhatsApp, and X (formerly Twitter), which have previously been shown to be effective for digital recruitment in health research.

Only those who provide consent will be enrolled in the study, in accordance with ethical guidelines for digital health research.

Sample Size Determination The sample size will be calculated using G*Power version 3.1, a well-established tool for statistical power analysis. Assuming a two-tailed independent samples t-test, an alpha level of 0.05, a power of 0.80, and a large effect size (Cohen's d = 0.83), the minimum required sample size will be 48 participants, with 24 participants per group. This sample size will provide sufficient power to detect large differences in asthma-related knowledge outcomes.

Randomization and Allocation Following informed consent, participants will be randomly assigned in a 1:1 ratio to either the intervention or control group. Randomization will be executed manually using a balloting technique, ensuring equal allocation and minimizing allocation bias. Due to the visible nature of the media intervention, participant blinding will not be possible, and the study will therefore adopt an open-label design.

Intervention Participants in the intervention arm will be asked to watch House M.D., Season 1, Episode 1, which includes dramatized depictions of asthma-related clinical scenarios. Prior research has demonstrated that medical TV dramas can enhance viewers' health literacy and influence decision-making, particularly in younger audiences. After viewing the episode, participants will complete a structured post-test questionnaire.

Participants in the control group will complete the same questionnaire at the same time intervals but will not view the media intervention. No additional educational content will be provided to either group during the study period.

Study Instruments The study instruments that will be used in this RCT are a pre-test and a post-test questionnaire. Both questionnaires will obtain, inter alia, data on the sociodemographic characteristics of the participants and their knowledge of asthma.

To ensure content validity, the initial draft of the questionnaire will be reviewed by two clinical experts in respiratory medicine. A pilot test involving five individuals (meeting the inclusion criteria but excluded from the trial) will be conducted to evaluate clarity, comprehension, and administration time. Feedback from the pilot will inform minor revisions to item structure and wording.

Participants in the intervention group will complete the questionnaire as a pre-test before viewing the episode and a post-test immediately afterward. Control group participants will complete the same questionnaire at matched time points without viewing the episode. Each correct answer will score one point, yielding a maximum score of 10. This outcome measure is focused exclusively on cognitive knowledge acquisition, and no secondary outcomes such as behavioral intent or media perception will be assessed.

Data will be collected using encrypted digital forms via Google Forms®. All responses will be time-stamped and automatically stored on password-protected institutional servers accessible only to the research team. Responses with more than 20% missing data will be excluded from analysis to ensure quality. Additional quality control procedures will include screening for contradictory answers, unusually fast completion times (e.g., under one minute), and potential duplicate submissions identified via IP and timestamp monitoring.

Statistical Analysis Descriptive statistics, including means, standard deviations, and frequencies, will be used to summarize participant demographics and outcome data. For inferential analysis, paired t-tests will be applied to assess within-group changes in knowledge scores (pre- vs. post-test), while independent samples t-tests will compare changes between the intervention and control groups. The Shapiro-Wilk test will be used to evaluate the normality of score distributions. When normality assumptions are violated, appropriate non-parametric tests such as the Wilcoxon signed-rank test and Mann-Whitney U test will be used. A p-value < 0.05 will be considered statistically significant.

Ethical Considerations Ethical approval has been obtained from the Institutional Review Board of Caleb University, Nigeria (CUL 25/0877). All participants will provide electronic informed consent before enrolment. They will be informed of their right to withdraw from the study at any time without penalty. All procedures will comply with international ethical standards for digital research involving human subjects.

Trial Timeline Participant recruitment and pre-test will be done in Weeks 2 and 3. The intervention will be administered in Week 4, and post-test will be done in Weeks 8 to 9. Data cleaning and analysis were conducted in Weeks 10 and 11, and the results will be compiled and disseminated in Weeks 12 to 16.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are between 18 and 35 years of age.
* Individuals who are proficient in English.
* Individuals who have access to a stable internet connection, a screen-enabled device, and Netflix movie platform.

Exclusion Criteria:

* Individuals with prior formal medical education.
* Individuals with a clinical history of asthma.
* Individuals who do not have access toa stable internet connection, a screen-enables device, or Netflix movie platform.
* Individuals who are aged below 18 years or above 35 years.
* Individuals who are concurrently participating in another asthma-related study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-04-25 (Estimated)

PRIMARY OUTCOMES:
Rate of change in asthma-related knowledge using questionnaire. | 5-months
  The rate of change in asthma-related knowledge assessed using a 10-item multiple-choice questionnaire developed specifically for this trial. Each item in the questionnaire will evaluate understanding of key asthma-related concepts featured in the TV drama, including symptoms, triggers, complications, medication, and clinical decision-making. This outcome measure is focused exclusively on cognitive knowledge acquisition.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. WHO Fact Sheet on asthma. Available online from https://www.who.int/. Accessed May 18, 2025. 2. Moris MJ. Asthma: practice, essentials, background, anatomy. Available online from https://emedicine.medscape.com/article/296301-overview#a1. Accessed May 18, 2025. 3. GBD 2021 Asthma and Allergic Diseases Collaborators. Global, regional, and national burden of asthma and atopic dermatitis, 1990-2021, and projections to 2050: a systematic analysis of the Global Burden of Disease Study 2021. Lancet Respir Med. 2025;13(5):425-446. doi:10.1016/S2213-2600(25)00003-7 4. Yuan L, Tao J, Wang J, et al. Global, regional, national burden of asthma from 1990 to 2021, with projections of incidence to 2050: a systematic analysis of the global burden of disease study 2021. eClinicalMedicine, Volume 80, 103051 5. Nunes C, Pereira AM & Morais-Almeida, M. Asthma costs and social impact. asthma res and pract . 2017;3(1). https://doi.org/10.1186/s40733-016-0029-3 6. Chan YY, Teh CH, Lim KK et al. Lifestyle, chronic diseases and self-rated health among Malaysian adults: results from the 2011 National Health and Morbidity Survey (NHMS). BMC Public Health. 2015;15(1). 7. Aneeshkumar S, Singh RB. Economic burden of asthma among patients visiting a private hospital in South India. Lung India. 2018 Jul-Aug;35(4):312-315. doi: 10.4103/lungindia.lungindia_474_17. 8. Ndarukwa P, Chimbari MJ & Sibanda EN. Development of a framework for increasing asthma awareness in Chitungwiza, Zimbabwe. asthma res and pract 5, 4 (2019). https://doi.org/10.1186/s40733-019-0052-2 9. Poureslami IM, Rootman I, Balka E, Devarakonda R, Hatch J, Fitzgerald JM. A systematic review of asthma and health literacy: a cultural-ethnic perspective in Canada. MedGenMed. 2007 Aug 21;9(3):40. 10. Basima A Almomani, Shoroq M Altawalbeh, Munther S Alnajjar, Suleiman M Momany, Assessment of medication knowledge among patients with asthma, Journal of Pharmaceutical Health Services Research, Volume 11, Issue 4, November 2020, Pages 349-354, https://doi.org/10.1111/jphs.12383 11. Basheti IA, Obeidat NM, Reddel HK. Inhaler technique education and asthma control among patients hospitalized for asthma in Jordan. Saudi Pharm J. 2018;26(8):1127-1136. doi:10.1016/j.jsps.2018.06.002 12. Dhruve H. Management of asthma: Adherence, inhaler technique and self-management. Practice Nursing 2018; 29: 4. 13. WHO 14. Orozco-Olvera V, Shen F, Cluver L. The effectiveness of using entertainment education narratives to promote safer sexual behaviors of youth: A meta-analysis, 1985-2017. PLoS One. 2019 Feb 12;14(2):e0209969. doi: 10.1371/journal.pone.0209969. 15. Francis A, Abraham E, Verma G, et al. (September 21, 2024) Assessment of Knowledge and Attitude of Asthmatic Patients and Their Caregivers Regarding the Disease Using an Asthma Knowledge Questionnaire in a Tertiary Care Hospital in Chennai. Cureus 16(9): e69832. doi:10.7759/cureus.69832